CLINICAL TRIAL: NCT01991808
Title: A Pilot Study to Assess the Suitability of DCE-MRI for Detection of Vascular Changes After Vaginal Brachytherapy
Brief Title: Suitability of DCE-MRI for Detection of Vascular Changes After VBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 26812
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Carcinoma of the Cervix, Carcinoma or Carcinosarcoma of the Uterus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCE-MRI (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy

SUMMARY:
This is a pilot study of DCE MR imaging to detect vascular changes in the vagina during and after radiotherapy n patients receiving adjuvant brachytherapyfor cervical or endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age.
* Must have histologically confirmed carcinoma of the cervix, carcinoma or carcinosarcoma of the uterus.
* Subjects are receiving intracavitary brachytherapy.
* ECOG performance status of 0-2.
* Creatinine clearance 30.

Exclusion Criteria:

* Subjects with an inability to tolerate MR imaging (i.e. claustrphobia)
* Study subjects who have contraindication to MRI scanning such as but not limited to subjects with pacemakers, metal fragments in the eye or certain metallic implants.
* Patients who do not speak or read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DCE-MRI: Radiotherapy and dynamic contrast enhanced magnetic resonance imaging
Period: Overall Study
Arm/Group | DCE-MRI
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DCE-MRI: Radiotherapy
Arm/Group | DCE-MRI
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | DCE-MRI
Number analyzed (Participants) | 16
Participants | 10

ADVERSE EVENTS:
Arm/Group | DCE-MRI
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DCE-MRI (N=16)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 1 (1)
Infection, Pelvis NOS (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Urethral pain (General disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes